CLINICAL TRIAL: NCT06893510
Title: The Effect of Virtual Reality-Based and Face-to-Face Relaxation Programs on Maternal and Fetal Outcomes in Pregnant Women With Preeclampsia
Brief Title: Virtual Reality-Based and Face-to-Face Relaxation Programs in Pregnant Women With Preeclampsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Güzin Ünlü Suvari, M.Sc, Ph.D. Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-01/37
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pre-Eclampsia; Maternal Health; Relaxation; Virtual Reality; Fetal Monitoring
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: This study follows a parallel-group design, where participants are randomly assigned to one of three independent groups: Face-to-Face Progressive Muscle Relaxation (F2F-PMRG), Virtual Reality Progressive Muscle Relaxation (VR-PMRG), or the Control Group.
Who Masked: Participant
Masking Description: This study employs a single-blind design, where participants will be unaware of their assigned intervention group (VR-based progressive muscle relaxation or in-person progressive muscle relaxation). However, researcher administering the interventions will be informed of group assignments. To ensure ethical compliance, separate informed consent forms have been prepared for each group, detailing the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-Face Progressive Muscle Relaxation Group (F2F-PMRG) (Experimental): Participants in this group will engage in 15-minute progressive muscle relaxation (PMR) exercises guided by the researcher for three consecutive days (once per day). To promote continued practice, participants will receive an audio recording of the PMR session, narrated by the researcher. After the initial three supervised sessions, they will be asked to listen to this recording twice a week and log their practice on a provided tracking sheet. The researcher will follow up with participants via phone calls to monitor compliance.
  Interventions: Other: Face-to-Face Progressive Muscle Relaxation
- Virtual Reality Progressive Muscle Relaxation Group (VR-PMRG) (Experimental): Participants will undergo 15-minute VR-assisted PMR sessions for three consecutive days (once per day) under the researcher's supervision. The VR sessions will include relaxing nature scenes combined with the researcher's PMR audio guidance. After the initial three sessions, participants will receive the same PMR audio recording and will be instructed to listen to it twice a week, logging their sessions. The researcher will conduct phone follow-ups to ensure adherence.
  Interventions: Other: Virtual Reality Based Progressive Muscle Relaxation
- Control Group (No Intervention): Participants in the control group will not receive any relaxation intervention and will continue their usual daily routines.

INTERVENTIONS:
Other: Virtual Reality Based Progressive Muscle Relaxation — Participants engage in progressive muscle relaxation exercises using a virtual reality headset that provides immersive visual and auditory relaxation content. Sessions are conducted under researcher supervision, followed by self-guided practice using an audio recording.
  Arms: Virtual Reality Progressive Muscle Relaxation Group (VR-PMRG)
Other: Face-to-Face Progressive Muscle Relaxation — Participants practice progressive muscle relaxation exercises in a traditional face-to-face setting, guided by a researcher. Initial supervised sessions are complemented by self-guided practice using an audio recording.
  Arms: Face-to-Face Progressive Muscle Relaxation Group (F2F-PMRG)

SUMMARY:
Preeclampsia, affecting 2-8% of pregnancies globally, is a leading hypertensive disorder in pregnancy. It is clinically characterized by elevated blood pressure (≥140/90 mmHg) after the 20th gestational week, often accompanied by proteinuria and systemic complications such as thrombocytopenia, liver dysfunction, and cerebral symptoms. This condition poses significant risks for both maternal and fetal health, increasing the likelihood of organ damage, preterm birth, and long-term cardiovascular and neurodevelopmental complications. Non-pharmacological interventions, including relaxation techniques, have been explored for symptom management. Progressive muscle relaxation (PMR) has shown efficacy in reducing stress, anxiety, and blood pressure. Recently, virtual reality (VR)-based relaxation techniques have gained attention for enhancing stress relief and improving health outcomes. This study aims to compare the effects of VR-based PMR with in-person PMR on maternal and fetal outcomes in preeclamptic pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with a diagnosis of preeclampsia.
* Gestational age ≥26 weeks.
* 18 years or older.
* Singleton and viable pregnancy.
* Willing to participate in the study voluntarily.

Exclusion Criteria:

* Multiple pregnancy.
* Pregnancy achieved through assisted reproductive technologies.
* Hearing or vision impairment in the pregnant individual.
* Fetal distress requiring emergency intervention.
* HELLP Syndrome or Eclampsia.
* History of vertigo.

Withdrawal Criteria:

* Cases where live birth does not occur.
* Participants who voluntarily withdraw from the study.
* Participants whose general health condition deteriorates during the intervention.
* Participants experiencing side effects from virtual reality headset use (e.g., dizziness, nausea, headache).
* Participants who do not practice progressive muscle relaxation at least once a week after the intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Descriptive Information Form | Day 1 (Baseline, Pre-Intervention)
  A researcher-developed questionnaire designed to collect sociodemographic and obstetric data based on the literature.
Maternal-Fetal Outcomes Follow-up Form | Day 1 (Baseline, Pre-Intervention), Day 2 and 3 (Post-Intervention for intervention groups, routine monitoring for the control group)
  Tracked using a researcher-developed follow-up form, including maternal vital signs and Non-Stress Test (NST) parameters.
Beck Anxiety Inventory (BAI) | Day 1 (Baseline, before intervention for intervention groups, before routine assessment for control group) and Day 3 (Post-intervention for intervention groups, after routine assessment for control group).
  Developed by Beck, Steer, Epstein, and Brown in 1988 and adapted into Turkish by Ulusoy et al. in 1998, this 21-item Likert-type scale measures anxiety levels. Each item is scored between 0 and 3, with total scores ranging from 0 to 63. Higher scores indicate higher levels of anxiety. The Turkish version has a Cronbach's alpha of 0.93, indicating high internal consistency. Factor analysis suggests two subscales: Subjective Symptoms and Somatic Symptoms.
Prenatal Comfort Scale (PCS) | Day 1 (Baseline, before intervention for intervention groups, before routine assessment for control group) and Day 3 (Post-intervention for intervention groups, after routine assessment for control group).
  Originally developed by Takeishi et al. in 2011 in Japan and later revised by Nakamura et al. in 2015 to a 15-item version, this scale measures prenatal comfort across five subscales: Partner's Role in Fatherhood, Fetal Interaction, Social Support, Maternal Role Adaptation, and Awareness of Pregnancy Changes. The 6-point Likert-type scale ranges from 0 (strongly disagree) to 5 (strongly agree), with higher scores indicating higher comfort levels. The scale has a Cronbach's alpha of 0.95 in the original study and 0.82 in the Turkish adaptation.
Heart Rate Variability (HRV) Measurement via Photoplethysmography (PPG) | Day 1 (Baseline, before the relaxation intervention) and Day 3 (Post-intervention, after the relaxation session).
  A non-invasive test used to assess physiological stress levels by measuring heart rate variability (HRV) through a photoplethysmography (PPG) sensor placed on the fingertip.
Satisfaction Evaluation Form (VAS) | Day 3 (Post-Intervention)
  A researcher-developed form assessing participants' overall satisfaction with the intervention, perceived anxiety and stress reduction, and general experience. (only for intervention groups)
Edinburgh Postpartum Depression Scale (EPDS) | Up to 4-6 weeks postpartum (via phone follow-up)
  eveloped by Cox et al. in 1987 and adapted into Turkish by Engindeniz et al. in 1996, this 10-item, 4-point Likert-type self-report scale assesses postpartum depression risk. Scores range from 0 to 30, with a cut-off point of 13. Internal consistency in the Turkish adaptation is 0.79, with a sensitivity of 0.84 and specificity of 0.88.
Postpartum Evaluation Form | Up to 4-6 weeks postpartum (via phone follow-up)
  A researcher-developed form assessing delivery type, maternal and neonatal health parameters, and newborn evaluations based on literature

CONTACTS AND LOCATIONS:
Overall Officials: Ergül Aslan, Prof. Dr., Principal Investigator — İstanbul University-Cerrahpaşa
Locations (1):
- Ümraniye Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be stored in an online database (e.g., Mendeley). Data will be available upon request after the study results are published by the researchers.

REFERENCES:
- [Background] Gestational Hypertension and Preeclampsia: ACOG Practice Bulletin, Number 222. Obstet Gynecol. 2020 Jun;135(6):e237-e260. doi: 10.1097/AOG.0000000000003891. PMID 32443079
- [Background] Bell IH, Nicholas J, Alvarez-Jimenez M, Thompson A, Valmaggia L. Virtual reality as a clinical tool in mental health research and practice . Dialogues Clin Neurosci. 2020 Jun;22(2):169-177. doi: 10.31887/DCNS.2020.22.2/lvalmaggia. PMID 32699517
- [Background] Bernstein, D. A., Borkovec, T. D., & Hazlett-Stevens, H. (2000). New directions in progressive relaxation training: A guidebook for helping professionals. Praeger Publishing.
- [Background] Chuang LL, Lin LC, Cheng PJ, Chen CH, Wu SC, Chang CL. The effectiveness of a relaxation training program for women with preterm labour on pregnancy outcomes: a controlled clinical trial. Int J Nurs Stud. 2012 Mar;49(3):257-64. doi: 10.1016/j.ijnurstu.2011.09.007. Epub 2011 Oct 2. PMID 21968280
- [Background] Dominguez-Solis E, Lima-Serrano M, Lima-Rodriguez JS. Non-pharmacological interventions to reduce anxiety in pregnancy, labour and postpartum: A systematic review. Midwifery. 2021 Nov;102:103126. doi: 10.1016/j.midw.2021.103126. Epub 2021 Aug 14. PMID 34464836
- [Background] Escobar-Bermudez A, Bejarano-Beltran MP. Experiences of women with preeclampsia in an Obstetric Intensive Care Unit in Colombia. Enferm Clin (Engl Ed). 2021 May-Jun;31(3):166-174. doi: 10.1016/j.enfcli.2020.11.003. Epub 2021 Jan 9. English, Spanish. PMID 33436348
- [Background] Estrella-Juarez F, Requena-Mullor M, Garcia-Gonzalez J, Lopez-Villen A, Alarcon-Rodriguez R. Effect of Virtual Reality and Music Therapy on the Physiologic Parameters of Pregnant Women and Fetuses and on Anxiety Levels: A Randomized Controlled Trial. J Midwifery Womens Health. 2023 Jan;68(1):35-43. doi: 10.1111/jmwh.13413. Epub 2022 Nov 16. PMID 36383473
- [Background] Ferguson C, Davidson PM, Scott PJ, Jackson D, Hickman LD. Augmented reality, virtual reality and gaming: an integral part of nursing. Contemp Nurse. 2015;51(1):1-4. doi: 10.1080/10376178.2015.1130360. Epub 2016 Jan 14. No abstract available. PMID 26678947
- [Background] Folk DM. Hypertensive Disorders of Pregnancy: Overview and Current Recommendations. J Midwifery Womens Health. 2018 May;63(3):289-300. doi: 10.1111/jmwh.12725. Epub 2018 May 15. PMID 29764001
- [Background] Hajesmaeel-Gohari S, Sarpourian F, Shafiei E. Virtual reality applications to assist pregnant women: a scoping review. BMC Pregnancy Childbirth. 2021 Mar 25;21(1):249. doi: 10.1186/s12884-021-03725-5. PMID 33765969
- [Background] Ioannou A, Papastavrou E, Avraamides MN, Charalambous A. Virtual Reality and Symptoms Management of Anxiety, Depression, Fatigue, and Pain: A Systematic Review. SAGE Open Nurs. 2020 Aug 27;6:2377960820936163. doi: 10.1177/2377960820936163. eCollection 2020 Jan-Dec. PMID 33415290
- [Background] Machado MSR, Bertagnolli TV, Veiga ECA, Ferreira CJH, Duarte G, Machado JSR, Carvalho R. Multiprofessional care promotes of quality of life in pregnant women with preeclampsia: a cross-sectional study. Clinics (Sao Paulo). 2020 Oct 26;75:e1951. doi: 10.6061/clinics/2020/e1951. eCollection 2020. PMID 33146357
- [Background] Severi FM, Prattichizzo D, Casarosa E, Barbagli F, Ferretti C, Altomare A, Vicino A, Petraglia F. Virtual fetal touch through a haptic interface decreases maternal anxiety and salivary cortisol. J Soc Gynecol Investig. 2005 Jan;12(1):37-40. doi: 10.1016/j.jsgi.2004.07.006. PMID 15629669
- [Background] Son H, Ross A, Mendoza-Tirado E, Lee LJ. Virtual Reality in Clinical Practice and Research: Viewpoint on Novel Applications for Nursing. JMIR Nurs. 2022 Mar 16;5(1):e34036. doi: 10.2196/34036. PMID 35293870